Title:

Explore the association of nonalcoholic fatty liver disease and atrial fibrillation in an elderly Chinese population

Date:

2017/12/3

Objective: Explore the association of nonalcoholic fatty liver disease and atrial fibrillation in an elderly Chinese population

Design: Compose a cross-sectional study analysing clinical data of the elderly adults ( $\geq$  65 years) who took health examination in Zhenhai Lianhua hospital, Ningbo, China in 2014.

## Methods:

- Get the approval of Hospital Ethics Committee for this study.
- Gather the physical examination results of the elderly adults (≥65 years old) who had undergone an annual physical examination at Zhenhai Lianhua Hospital, Ningbo, China in 2014.
- Exclude the following participants: (1) those with unknown alcohol intake or excessive alcohol intake; (2) those with unknown BMI or BMI ≤ 18.0kg/m2; (3) those with incomplete basic physical data; (3) those with missing liver ultrasonic diagnosis; (4) those with unknown causes of chronic liver disease.
- Verbally informe all the participants and get agreement to participate in the study.
- Analyse the physical examination results of the participants using Student's t-test or the Mann-Whitney U test or chi-square test or Fisher's exact test.
- Make tables and charts.
- Analyse the results and write paper.